CLINICAL TRIAL: NCT00377455
Title: Placebo Controlled Trial of Bosentan vs Placebo in NYHA Class I/II Scleroderma Patients With Exercise Induced Pulmonary Hypertension
Brief Title: Placebo Controlled Trial of Bosentan in Scleroderma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to inadequate enrolment
Sponsor: Georgetown University (Other)
Collaborators: Actelion (Industry)
Responsible Party: Principal Investigator, Virginia Steen, MD, Professor of Medicine, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 06-043; Bosentan (Other: Georgetown University)
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Results first posted 2011-07-20 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-04

CONDITIONS: Systemic Scleroderma; Pulmonary Hypertension
Keywords: scleroderma; systemic sclerosis; bosentan; pulmonary hypertension; PHAROS; PHROS; exercise echocardiogram
MeSH Terms: conditions — Scleroderma, Systemic; Hypertension, Pulmonary; Scleroderma, Diffuse | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bosentan (Experimental)
  Interventions: Drug: Bosentan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosentan — 62.5 mg by mouth (PO) twice daily (Bid) for 1 month, followed by 125 mg PO Bid thereafter, for a total of 16 weeks
  Arms: Bosentan
Drug: Placebo — 62.5 mg PO Bid for 1 month, followed by 125 mg PO Bid thereafter, for a total of 16 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the drug Bosentan improves exercise tolerance in scleroderma patients.

DETAILED DESCRIPTION:
Pulmonary hypertension (PAH) is a common and usually fatal form of lung disease in systemic sclerosis (SSc). Multiple drugs have been approved for the treatment of New York Heart Association (NYHA)Class III/IV PAH in scleroderma. Bosentan is an endothelin-1 antagonist which showed significant improvement in distance walked during 12 week clinical trials in PAH patients (7). Therapy for asymptomatic systemic sclerosis patients diagnosed incidentally with PAH (World Health Organization (WHO) Functional Class I) remains controversial. We hypothesize that asymptomatic or minimally symptomatic patients with systemic sclerosis and normal resting pulmonary artery pressures who demonstrate an abnormal rise in pulmonary artery systolic pressure with stress Doppler echocardiography testing represent a subset of patients who already have pulmonary vascular disease and who are at risk for the development of severe PAH. We further hypothesize that early identification and treatment of such patients may retard the progression of that disease.

Hypotheses:

1. Stress echocardiography identifies early pulmonary vascular disease by detecting exercise-induced pulmonary hypertension in patients with systemic sclerosis.
2. Treatment of exercise-induced PAH with Bosentan will lead to improved exercise endurance in patients with systemic sclerosis.

Subjects will be recruited from those patients who have had an abnormal exercise test as part of an earlier study, Exercise Echocardiograms in Scleroderma (IRB# 03-363).

ELIGIBILITY:
Inclusion Criteria:

* SSc patients > 18 with NYHA functional Class I/II symptoms, informed consent, and who are willing to participate in the Pulmonary Hypertension Assessment and Recognition of Outcomes in Scleroderma (PHAROS) long term study (Georgetown IRB 04-227)
* Right heart catheterization with

  1. Normal Mean Pulmonary Arterial Pressure (PAP) at rest
  2. Mean PAP > 30 with exercise
  3. Wedge Pressure < 18
* Entry criteria for participating in the exercise echocardiogram study (Georegtown IRB 03-363)

  1. Diffusing Capacity (DLCO) <60 with a Forced Vital Capacity (FVC) >60%, or
  2. FVC/DLCO > 1.6, or
  3. a resting Pulmonary Arterial Systolic Pressure (PASP)> 40mmHg

Exclusion Criteria:

* Established resting pulmonary hypertension
* Congestive heart failure
* Diastolic dysfunction
* Pregnancy
* Inability to adequately walk/exercise
* Severe liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia D Steen, MD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - University of Connecticut, Farmington, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia

REFERENCES:
- [Background] Stupi AM, Steen VD, Owens GR, Barnes EL, Rodnan GP, Medsger TA Jr. Pulmonary hypertension in the CREST syndrome variant of systemic sclerosis. Arthritis Rheum. 1986 Apr;29(4):515-24. doi: 10.1002/art.1780290409. PMID 3707629
- [Background] Yousem SA. The pulmonary pathologic manifestations of the CREST syndrome. Hum Pathol. 1990 May;21(5):467-74. doi: 10.1016/0046-8177(90)90002-m. PMID 2186993
- [Background] al-Sabbagh MR, Steen VD, Zee BC, Nalesnik M, Trostle DC, Bedetti CD, Medsger TA Jr. Pulmonary arterial histology and morphometry in systemic sclerosis: a case-control autopsy study. J Rheumatol. 1989 Aug;16(8):1038-42. PMID 2585400
- [Background] MacGregor AJ, Canavan R, Knight C, Denton CP, Davar J, Coghlan J, Black CM. Pulmonary hypertension in systemic sclerosis: risk factors for progression and consequences for survival. Rheumatology (Oxford). 2001 Apr;40(4):453-9. doi: 10.1093/rheumatology/40.4.453. PMID 11312386
- [Background] Grunig E, Janssen B, Mereles D, Barth U, Borst MM, Vogt IR, Fischer C, Olschewski H, Kuecherer HF, Kubler W. Abnormal pulmonary artery pressure response in asymptomatic carriers of primary pulmonary hypertension gene. Circulation. 2000 Sep 5;102(10):1145-50. doi: 10.1161/01.cir.102.10.1145. PMID 10973844
- [Background] Steen V, Medsger TA Jr. Predictors of isolated pulmonary hypertension in patients with systemic sclerosis and limited cutaneous involvement. Arthritis Rheum. 2003 Feb;48(2):516-22. doi: 10.1002/art.10775. PMID 12571862
- [Background] Rubin LJ, Badesch DB, Barst RJ, Galie N, Black CM, Keogh A, Pulido T, Frost A, Roux S, Leconte I, Landzberg M, Simonneau G. Bosentan therapy for pulmonary arterial hypertension. N Engl J Med. 2002 Mar 21;346(12):896-903. doi: 10.1056/NEJMoa012212. PMID 11907289

RESULTS

PARTICIPANT FLOW:
Groups:
- Bosentan and Placebo Arms: This group consists of subjects on both arms of the study - bosentan and placebo
Period: Overall Study
Arm/Group | Bosentan and Placebo Arms
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bosentan and Placebo Arms
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Exercise Time on the Exercise Echocardiogram Using the Standard Bruce Stress Protocol.
Description: The total exercise time measured using the exercise echocardiogram is evaluated with the standard Bruce Stress Protocol, and this will be determined after 16 weeks on the study medication.
Time Frame: This will be determined after 16 weeks on the study medication.
Groups:
- Bosentan/Placebo: Outcomes not available, due to early termination of study
Arm/Group | Bosentan/Placebo
Number analyzed (Participants) | 0

2. Secondary Outcome: 6-minute Walk Distance
Description: The distance walked during a 6-minute walk test.
Time Frame: 16 weeks
Population: Outcomes not available, due to early termination of study
Arm/Group | Bosentan/Placebo
Number analyzed (Participants) | 0

3. Secondary Outcome: Brain Natriuretic Peptide (BNP) Level
Description: Serum BNP level to evaluate Brain Natriuretic Peptide (BNP) level
Time Frame: 16 weeks
Population: Outcomes not available, due to early termination of study
Arm/Group | Bosentan/Placebo
Number analyzed (Participants) | 0

4. Secondary Outcome: Endothelin-1(ET-1) Level
Description: From saved serum to determine Endothelian-1 (ET-1) levels in patients
Time Frame: 16 weeks
Population: Outcomes not available, due to early termination of study
Arm/Group | Bosentan/Placebo
Number analyzed (Participants) | 0

5. Secondary Outcome: Quality of Life (QOL)
Description: QOL is measured using the Short Form 36 Health Survey (SF-36, which measures health on eight dimensions: general health perception, physical and social functioning, role limitations by physical or emotional problems, mental health, vitality, and bodily pain. For each dimension items are coded, summed, and transformed on to a scale from 0 (worst health) to 100 (best health).
Time Frame: 16 weeks
Population: Outcomes not available, due to early termination of study
Arm/Group | Bosentan/Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Serious or Other (non-serious) Adverse Events were collected/assessed, but none observed
Arm/Group | Bosentan and Placebo Arms
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No